CLINICAL TRIAL: NCT00354328
Title: Relationship of Diastolic Function and Functional Capacity in Hypertrophic Cardiomyopathy: A Post-Hoc Analysis of Protocols 01-H-0066 and 96-H-0144
Brief Title: Heart Function and Exercise Capacity in Patients With Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050163; 05-H-0163
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2017-10

CONDITIONS: Angina, Unstable; Myocardial Infarction; Ischemic Heart Disease
Keywords: HCM; Echocardiography; Diastolic Dysfunction; Enalapril
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction; Myocardial Ischemia

SUMMARY:
This study will examine the relationship between certain measures of heart function and exercise capacity in patients with hypertrophic cardiomyopathy (HCM).

Patients who participated in NHLBI studies 01-H-0006 ("Double Blind Placebo-Controlled Study of Pirfenidone - A Novel Anti-Fibrotic Drug - in Symptomatic Patients with Hypertrophic Cardiomyopathy Associated with Left Ventricular Diastolic Dysfunction") and 96-H-0144 ("Double Blind Placebo-Controlled Study of Long-Term Effects of Angiotensin-Converting Enzyme Inhibition (Enalapril) and Angiotensin II Receptor Blockade (Losartan) on Genetically-Induced Left Ventricular Diastolic Dysfunction") are eligible for this study. Data from echocardiograms and measures of left ventricular pressure obtained from patients in those studies will be analyzed in the current study to assess their influence on exercise capacity. No additional tests, treatments or other procedures are required.

Information from this study may help in the development of improved drug treatments for HCM.

DETAILED DESCRIPTION:
NIH Protocols 01-H-0066, Double Blind Placebo Controlled Study of Pirfenidone A Novel Anti-Fibrotic Drug in Symptomatic patients with Hypertrophic Cardiomyopathy (HCM) Associated with left Ventricular Diastolic Dysfunction and 96-H-0144, Double Blind Placebo-Controlled Study of Long-Term Effects of Angiotensin Converting Enzyme Inhibition (Enalapril) and Angiotensin II Receptor Blockade (Losartan) On Genetically-Induced Left Ventricular Diastolic Dysfunction were undertaken to assess the effect of therapeutic interventions on left ventricular (LV) diastolic function. The relationship between baseline measures of diastolic function as assessed by noninvasive modalities such as Doppler echocardiography and radionuclide angiography, and qualitative and objective measures of functional capacity in patients without LV outflow tract obstruction has not been reported. In this protocol we will look at measures of LV geometry, relaxation and novel indices of ventricular compliance as they may influence measures of exercise capacity. In all cases, we will use pre-existing baseline data obtained with informed consent as part of the above protocols.

ELIGIBILITY:
* Eligibility criteria not listed; Analysis of data from previous studies.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-05-27; Study Completion 2013-10-22

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea R McAreavey, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States